CLINICAL TRIAL: NCT04344418
Title: Impact of Nurse-Led Focused Cardiac Ultrasound Versus Usual Care on Time to Diagnosis in Adults With Cardiorespiratory Failure: A Two-Cluster Stepped Wedge Clinical Feasibility Trial
Brief Title: Harnessing Alternative Resources to Aid Kenyans With Acute Illness
Acronym: HARAKA-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: University of Oxford (Other); Kenyatta National Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Wangari Waweru-Siika, Assistant Professor, Aga Khan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 31-20
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Cardiorespiratory Failure

STUDY DESIGN:
Intervention Model Description: 2-cluster stepped wedge clinical feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): The control arm will consist of usual care ie a combination of physical examination, lab tests and imaging. The need for a formal echocardiographic evaluation by a cardiologist or cardiac sonographer in patients assigned to the control arm will be at the discretion of the clinical teams, as is usual care at the Kenyatta National Hospital (KNH) and Aga Khan University Hospital Nairobi (AKUHN). A diagnosis will be selected based on the same pre-defined checklist and the time the diagnosis is made recorded.
  Interventions: Other: Usual care
- Nurse-performed focused cardiac ultrasound (FoCUS) (Experimental): The experimental arm will consist of nurse-performed FoCUS for patients with cardiorespiratory failure. A FoCUS-trained nurse will perform a FoCUS examination within 30 minutes of triage by the triage clinician. The Philips Lumify® handheld ultrasound device (HUD) with a phased array probe will be used and studies limited to a maximum of 10 minutes each. A presumptive diagnosis will then be selected by the nurse from a FoCUS checklist based on pre-defined thresholds for each FoCUS target condition and the time the diagnosis is made recorded. Additional imaging and lab tests may be requested at the discretion of the clinical team but the FoCUS nurses will be blinded to the results of these.
  Interventions: Device: Nurse-performed Focused cardiac ultrasound (FoCUS)

INTERVENTIONS:
Device: Nurse-performed Focused cardiac ultrasound (FoCUS) — A FoCUS-trained nurse will perform a FoCUS examination within 30 minutes of triage by the triage clinician. The Philips Lumify® handheld ultrasound device (HUD) with a phased array probe will be used and studies limited to a maximum of 10 minutes each. A presumptive diagnosis will then be selected by the nurse from a FoCUS checklist based on pre-defined thresholds for each FoCUS target condition and the time the diagnosis is made recorded. Additional imaging and lab tests may be requested at the discretion of the clinical team but the FoCUS nurses will be blinded to the results of these.
  Arms: Nurse-performed focused cardiac ultrasound (FoCUS)
Other: Usual care — The control arm will consist of usual care ie a combination of physical examination, lab tests and imaging. The need for a formal echocardiographic evaluation by a cardiologist or cardiac sonographer in patients assigned to the control arm will be at the discretion of the clinical teams, as is usual care at KNH and AKUHN
  Arms: Usual care

SUMMARY:
Kenya does not have enough experts to perform heart scans in patients who are very sick and in need of urgent intervention. The purpose of this research is to find out whether training Kenyan nurses to perform basic heart scans would shorten the time it takes to know whether the heart and lungs are working normally in very sick patients, to guide treatment. Patients will be placed into one of two groups: One group will have a quick scan of the heart and lungs carried out by trained nurses to see how well these organs are working, in addition to receiving the normal care offered at the hospital. The other group will receive the normal care offered in the hospital only and will not have a scan performed by these nurses. The time it takes to make a diagnosis between the two groups will then be compared. Should the group that has heart scans by nurses be found to spend less time waiting for a diagnosis to be made, more nurses in Kenya will be trained to provide this service, to minimise delays in our emergency departments.

DETAILED DESCRIPTION:
Echocardiography is a useful, non-invasive diagnostic tool in time-critical emergencies. A national shortage of cardiologists and of doctors in Kenya however further compounds the problem of insufficient staff for emergency care and of any capacity building efforts. To achieve the goals of Sustainable Development Goal Number 3 (SDG-3) and realise the government's vision of universal healthcare for all, alternatives to the human resource challenge are key. Modifying the Scope of Practice of Kenyan nurses is one possible solution. Task-shifting traditionally cardiologist roles such as focused cardiac ultrasound (FoCUS) could shorten the time it takes to make a diagnosis in patients with cardiorespiratory failure of likely cardiac origin, making prolonged turnaround times in our public facilities a thing of the past. Our overarching aim is to harness the power of nurses doing FoCUS. The central hypothesis of this work is that in patients with cardiorespiratory failure, a nurse-led FoCUS-guided service would shorten time to diagnosis, supporting interventions and improving outcomes among the critically ill. Insight into potential barriers and enablers for the implementation of a nurse-performed FoCUS service in Kenya is crucial for the success of such a service redesign.

ELIGIBILITY:
Inclusion Criteria:

Any one of:

* Systolic blood pressure <90 millimetres of mercury (mmHg)
* Mean arterial pressure (MAP)<65 millimetres of mercury (mmHg)
* Shock index >1 (heart rate/systolic blood pressure)
* Respiratory rate > 30 breaths/minute
* Oxygen saturations <94%
* Arterial oxygen partial pressure (paO2) <60 millimetres of mercury (mmHg)
* Arterial carbon dioxide partial pressure (paCO2) >50 millimetres of mercury(mmHg)

Exclusion Criteria:

* Trauma
* Pregnancy
* Patients requiring immediate life-saving interventions eg cardiopulmonary resuscitation (CPR) or defibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis | 24 hours
  Difference in median time to diagnosis between nurse-performed FoCUS and usual care.

SECONDARY OUTCOMES:
Number of patients with cardiorespiratory failure who have a FoCUS exam performed in A&E | 10 months
  Number of patients with cardiorespiratory failure who have a FoCUS
Proportion of patients with cardiorespiratory failure who have a FoCUS exam performed in A&E | 10 months
  Proportion of patients with cardiorespiratory failure who have a FoCUS
Diagnostic accuracy of nurse-performed FoCUS | 10 months
  Sensitivity and specificity of novice FoCUS compared to a reference standard (cardiologist opinion)
Number of FoCUS protocol components suitable for inclusion in a local FoCUS curriculum | 10 months
  Number of FoCUS protocol components suitable for inclusion in a local FoCUS curriculum
Proportion of novice scanners able to access remote supervision for FoCUS practice. | 10 months
  Proportion of novice scanners able to access remote supervision for FoCUS practice.

CONTACTS AND LOCATIONS:
Overall Officials: Wangari Waweru-Siika, FRCA, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: Yes
Available on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Available on request